CLINICAL TRIAL: NCT02134262
Title: Clinical Research of Gene Therapy for Refractory B-Cell Non-Hodgkin Lymphoma Using Autologous T Cells Expressing a Chimeric Antigen Receptor Specific to the CD19 Antigen
Brief Title: Gene Therapy for B-Cell Non-Hodgkin Lymphoma Using CD19 CAR Gene Transduced T Lymphocytes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jichi Medical University (Other)
Collaborators: Takara Bio Inc. (Industry)
Responsible Party: Principal Investigator, Keiya Ozawa, Professor, Jichi Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JMU-CD19CAR
Record Dates: First submitted 2014-04-16; First posted 2014-05-09 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Keywords: Anti-CD19 CAR Expressing T cells Therapy; CD19 CAR Gene-Transduced Lymphocyte; Adoptive Immunotherapy; Genetically Engineered Lymphocyte Therapy; Retroviral Vector; Burkitt Lymphoma; Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphomatoid Granulomatosis; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Mantle-Cell; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Experimental; Immune System Diseases
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphomatoid Granulomatosis; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Mantle-Cell; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Experimental; Immune System Diseases | interventions — Cyclophosphamide; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level -1 (Experimental): Cyclophosphamide or Bendamustine as Pre-treatment, and in combination with CD19-CAR-T. In case when sufficient cell number of CD19-CAR-T has been manufactured, the physician judges whether the 2nd infusion of CD19-CAR-T should be performed based on the condition of the subject.
  Interventions: Drug: Cyclophosphamide or Bendamustine; Genetic: Dose Level -1
- Dose Level 1 (Experimental): Cyclophosphamide or Bendamustine as Pre-treatment, and in combination with CD19-CAR-T. In case when sufficient cell number of CD19-CAR-T has been manufactured, the physician judges whether the 2nd infusion of CD19-CAR-T should be performed based on the condition of the subject.
  Interventions: Drug: Cyclophosphamide or Bendamustine; Genetic: Dose Level 1
- Dose Level 2 (Experimental): Cyclophosphamide or Bendamustine as Pre-treatment, and in combination with CD19-CAR-T. In case when sufficient cell number of CD19-CAR-T has been manufactured, the physician judges whether the 2nd infusion of CD19-CAR-T should be performed based on the condition of the subject.
  Interventions: Drug: Cyclophosphamide or Bendamustine; Genetic: Dose Level 2
- Dose Level 3 (Experimental): Cyclophosphamide or Bendamustine as Pre-treatment, and in combination with CD19-CAR-T. In case when sufficient cell number of CD19-CAR-T has been manufactured, the physician judges whether the 2nd infusion of CD19-CAR-T should be performed based on the condition of the subject.
  Interventions: Drug: Cyclophosphamide or Bendamustine; Genetic: Dose Level 3

INTERVENTIONS:
Drug: Cyclophosphamide or Bendamustine — Cyclophosphamide [1.5 g/m^2 x 1 day Intravenous (IV)] or Bendamustine [120 mg/m^2 x 2 days Intravenous (IV)] is administered as Pre-treatment medication of CD19-CAR-T.
Genetic: Dose Level -1 — CD19-CAR-T [1 x 10^5 cells/kg x 1 day and 2 x 10^5 cells/kg x 1 day Intravenous (IV)] are administered.
  Arms: Dose Level -1
Genetic: Dose Level 1 — CD19-CAR-T [1/3 x 10^6 cells/kg x 1 day and 2/3 x 10^6 cells/kg x 1 day Intravenous (IV)] are administered.
  Arms: Dose Level 1
Genetic: Dose Level 2 — CD19-CAR-T [1 x 10^6 cells/kg x 1 day and 2 x 10^6 cells/kg x 1 day Intravenous (IV)] are administered.
  Arms: Dose Level 2
Genetic: Dose Level 3 — CD19-CAR-T [1/3 x 10^7 cells/kg x 1 day and 2/3 x 10^7 cells/kg x 1 day Intravenous (IV)] are administered.
  Arms: Dose Level 3

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and blood kinetics of autologous T cells genetically modified to express anti-CD19 Chimeric Antigen Receptor in patients with relapsed or refractory B-Cell Non-Hodgkin Lymphoma.

DETAILED DESCRIPTION:
Peripheral blood (up to 600 mL) will be collected from a subject after obtaining a written informed consent and completing the 1st registration. Peripheral blood mononuclear cells (PBMCs) and plasma are obtained from the blood, and T cells contained in the PBMCs are transduced with anti-CD19 CAR gene by using SFG-1928z retroviral vector. Anti-CD19 CAR expressing T cells (CD19-CAR-T) will be expanded using a medium containing autologous plasma. After the T cells pass in quality control tests, the subject will go into 2nd registration. Subjects will be hospitalized and administered Cyclophosphamide on Day -2 or Bendamustine on Day -3 to Day -2 intravenously as Pre-treatment, and then subjects will receive 1st infusion of CD19-CAR-T on Day 0 and Day 1 (Day 1：1/3 dose, Day 2：2/3 dose) as a split dose. In case the sufficient cell number of CD19-CAR-T is manufactured, DLT is not observed after CD19-CAR-T infusion, certain clinical effect is observed and additional treatment is preferable, the necessity of 2nd infusion will be assessed. In the case that 2nd infusion is necessary, it is allowed to infuse at appropriate timing.

This study is conducted based on the 3+3 dose escalation scheme. Three subjects are enrolled in each group of Dose Level. If one of the 3 subjects show DLT during DLT assessment period, another 3 subjects will be added; therefore, decision as to whether the next Dose Level can follow or not is made based on the results obtained from the total of 6 subjects.

The investigator assesses the tumor shrinkage effect of CD19-CAR-T in accordance with "Revised response criteria malignant lymphoma", at 12 week after the 1st infusion of CD19-CAR-T (or at the time of termination). The investigator also assesses the safety during the follow-up period. Long-term follow-up study is conducted at frequency of once a year for 15 years after the 1st infusion of CD19-CAR-T in reference to guidelines of FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory B-NHL.
2. Evaluable region can be identified by CT scan and is positive by FDG-PET.
3. 20 ≤ age ≤ 70 years at the time of informed consent.
4. ECOG performance status of 0-2.
5. Well preserved main organ functions.
6. Life expectancy ≥3 months after informed consent.
7. Written informed consent.

Exclusion Criteria:

1. Other active malignancy.
2. CNS infiltration of lymphoma.
3. History of allogeneic stem cell transplantation.
4. Already participated in a clinical trial in which CD19-CAR-T are administered within 24 weeks.
5. Concurrent use of systemic steroids or immunosuppressive agents.
6. Concurrent severe heart disease.
7. History of severe cerebrovascular disease or sequela including paralysis.
8. Known active or severe infection.
9. HIV seropositive status.
10. HBsAg-positive or both HBcAb and HBV-DNA positive.
11. Active hepatitis C.
12. Psychiatric disorder or drug addiction that affects the ability of informed consent.
13. Pregnant or breastfeeding women, women who may be pregnant and women desiring to become pregnant. Men who desire impregnating a woman are also excluded (excluded: in case when sperm is cryopreserved prior to gene therapy and a child is born by using the sperm).
14. Any other patients judged by the investigators to be inappropriate for the subject of this study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity Profile | 12 weeks
  Confirm the toxicity profile with CTCAE ver4.0.
Toxicity Profile | 12 weeks
  Confirm existence or non-existence of normal B-lymphocytes decrease by flow cytometry.
Toxicity Profile | 12 weeks
  Measure immunoglobulin by PCR.
Toxicity Profile | 12 weeks
  Confirm replication competent retrovirus (RCR) by PCR.
Toxicity Profile | 12 weeks
  Confirm clonality by linear amplification mediated (LAM)-PCR.
Quality test of CD19-CAR-T | Before administration
  Transduction efficiency, viability, sterility and potency.

SECONDARY OUTCOMES:
Tumor shrinkage effect | 12 weeks
  Confirm the efficacy with "Revised response criteria for malignant lymphoma" J Clin Oncol. 25: 579-586 (2007).
Lymphocyte subset analysis of CD19-CAR-T | 12 weeks
  Confirm the state of immune mechanism by flow cytometry.
Human anti-mouse antibody (HAMA) test | 12 weeks
  Examine HAMA with ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Keiya Ozawa, MD, PhD, Study Chair — Division of Hematology, Department of Medicine, Center for Molecular Medicine, Division of Genetic Therapeutics, Center for Molecular Medicine, Division of Immuno-Gene & Cell Therapy (Takara Bio), Jichi Medical University
Locations (1):
- Jichi Medical University, Shimotsuke, Tochigi, Japan